CLINICAL TRIAL: NCT04497597
Title: Upadacitinib Treatment Patterns, Achievement of Treatment Targets and Maintenance of Response in Moderate to Severe Rheumatoid Arthritis Patients in Real-World Practice (UPHOLD)
Brief Title: A Study of Oral Upadacitinib Tablets to Assess Treatment Patterns, Achievement of Treatment Targets and Maintenance of Response in Adult Participants With Moderate to Severe Rheumatoid Arthritis
Acronym: UPHOLD
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-095
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Upadacitinib; RINVOQ
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving Upadacitinib: Participants receiving Upadacitinib for moderate to severe rheumatoid arthritis (RA).

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory disease of the joints causing pain, stiffness, swelling and loss of joint function. Despite the range of treatment options for RA steadily increasing, many patients remain sub-optimally managed, with sustained clinical remission rarely achieved. This study will assess the treatment patterns, achievement of treatment targets and maintenance of response.

Upadacitinib is a drug approved for the treatment of moderately to severely active rheumatoid arthritis. Adult participants with moderate to severe RA who have been prescribed upadacitinib by their physicians will be enrolled. Approximately, 1660 participants will be enrolled this study, worldwide.

Participants will not receive Upadacitinib as part of this study, but will be followed for response to treatment for up to 24 months.

There may be higher burden for participants in this trial compared to their standard of care. Participants will attend regular visits, every 3 months, during the course of the study at a hospital or clinic and will be asked to provide additional information by questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe active Rheumatoid Arthritis (RA).
* Physician decision on patient treatment with upadacitinib must have been reached prior to and independently of recruitment in the study.
* Upadacitinib prescribed in accordance to the applicable approved label and local regulatory and reimbursement policies.
* French Participants Only: Taking oral glucocorticoids ≥5 mg/day of prednisone or equivalent for at least 3 months prior to study start.

Exclusion Criteria:

- Prior treatment with Upadacitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving Upadacitinib according to the product prescribing information, for moderate to severe active Rheumatoid Arthritis (RA).
Sampling Method: Non-Probability Sample
Enrollment: 1532 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve Remission | At Month 6
  Remission is defined as Disease Activity Score at 28 joints (DAS28) C-reactive Protein (CRP)<2.6.
Percentage of Participants Who Achieve Remission at 6 Months and Maintain Remission | At Month 12
  Remission is defined as DAS28-CRP<2.6. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve Remission at 6 Months and Maintain Remission | At Month 24
  Remission is defined as DAS28-CRP<2.6. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.
Percentage of Participants Who Achieve Low Disease Activity (LDA) at 6 months that maintain LDA | Through Month 24
  LDA is defined as DAS28-CRP≤3.2. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.
Percentage of Participants Who Achieve Remission at 3 Months and Maintain Remission | Through Month 24
  Remission is defined as DAS28-CRP<2.6. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.
Percentage of Participants Who Achieve Remission at 6 Months and Maintain Remission Grouped by Glucocorticoid Dose | At Month 12
  Remission is defined as DAS28-CRP<2.6. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.
Percentage of Participants Who Achieve LDA at 3 months that maintain LDA Grouped by Glucocorticoid Dose | Through Month 6
  LDA is defined as DAS28-CRP≤3.2. Maintaining remission is defined as no more than 0.6 point increase in DAS28-CRP.
Percentage of Participants in LDA that Achieve Glucocorticoid Dose <5 mg/Day Per Visit | Through Month 24
  LDA is defined as DAS28-CRP<3.2.
Percentage of Participants in Remission that Achieve Glucocorticoid Dose <5 mg/Day Per Visit | Through Month 24
  Remission is defined as DAS28-CRP<2.6.
Percentage of Participants Who Achieved a Glucocorticoid Dose <5 mg/Day Without Conventional Synthetic Disease Modifying Anti Rheumatic Drug (csDMARD) Intensification | At Month 6
  Percentage of participants who achieved a glucocorticoid dose <5 mg/day without csDMARD intensification.
Percentage of Participants Who Initiated Upadacitinib as Combination Therapy (csDMARD +/- Glucocorticoids) That Moved to Monotherapy (+/- Glucocorticoids) | Through Week 24
  Percentage of participants who initiated Upadacitinib as combination therapy (csDMARD +/- Glucocorticoids) that moved to monotherapy (+/- glucocorticoids).
Of the Participants Initiating Upadacitinib as Combination Therapy (csDMARD +/- Glucocorticoids) and Achieve Remission at 6 months, the Percentage of Participants that Maintain Remission Grouped by Maintenance of Combination Therapy Strategy | Through Month 24
  Remission is defined as DAS28-CRP<2.6.
Of the Participants Initiating Upadacitinib as Combination Therapy (csDMARD +/- Glucocorticoids) and Achieve LDA at 6 months, the Percentage of Participants that Maintain LDA Grouped by Maintenance of Combination Therapy Strategy | Through Month 24
  LDA is defined as DAS28-CRP<3.2.
Of the Participants Initiating Upadacitinib as Monotherapy Therapy (+/- Glucocorticoids) and Achieve Remission at 6 months, the Percentage of Participants that Maintain Remission Grouped by Maintenance of Monotherapy | Through Month 24
  Remission is defined as DAS28-CRP<2.6.
Of the Participants Initiating Upadacitinib as Monotherapy Therapy (+/- Glucocorticoids) and Achieve LDA at 6 months, the Percentage of Participants that Maintain LDA Grouped by Maintenance of Monotherapy | Through Month 24
  LDA is defined as DAS28-CRP<3.2.
Percentage of Participants Who Do Not Achieve Remission at Any Point in the Study | Through Month 24
  Remission is defined as DAS28-CRP<2.6.
Time to the Discontinuation of Upadacitinib | Through Month 24
  Time to the discontinuation of Upadacitinib.
Time to First Treatment Adjustment | Baseline (Month 0) Through Month 24
  Treatment Adjustment is defined as treatment escalation/de-escalation/ addition/withdrawal.
Percentage of Participants Achieving LDA Grouped by Therapy Strategy | Through Month 24
  LDA is defined as DAS28-CRP<3.2, Simplified Disease Activity Index (SDAI) ≤11 and Clinical Disease Activity Index (CDAI) ≤10.
Percentage of Participants Achieving Remission Grouped by Therapy Strategy | Through Month 24
  Remission is defined as DAS28-CRP<2.6, SDAI≤3.3 and CDAI ≤2.8.
Change in Medication Burden Treatment Burden Questionnaire (TBQ) in Participants, Grouped by Therapy Strategy | Through Week 24
  The TBQ is composed of 13 items rated on a Likert scale ranging from 0 (not a problem), to 10 (big problem). scores can be summed into a global score, ranging from 0 to 130.
Change in Physical Function Health Assessment Questionnaire - Disability Index (HAQ-DI) in Participants, Grouped by Therapy Strategy | Baseline (Month 0) Through Month 24
  HAQ is a widely accepted, validated, rheumatology specific instrument to assess physical function in Rheumatoid Arthritis. It consists of 20 questions, covering eight types of activities. For each question, scores range from 0 to 3 (0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty or with assistance; 3 = unable to do). HAQ Disability Index (HAQ-DI) score is the average of the highest score in each of the eight categories.
Change in Pain Visual Analogue Scale (VAS) in participants, Grouped by Therapy Strategy | Baseline (Month 0) Through Month 24
  A VAS is used to assess worst joint pain in the past 7 days.
Change in Morning Stiffness in Participants, Grouped by Therapy Strategy | Baseline (Month 0) Through Month 24
  A numeric rating scale (NRS) is used to assess severity and length of morning stiffness in the past 7 days.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) in Participants, Grouped by Therapy Strategy | Baseline (Month 0) Through Month 24
  The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (0 = not at all fatigued to 4 = very much fatigued).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (263):
- Argentina (9):
  - Hospital Italiano La Plata /ID# 222190, La Plata, Buenos Aires
  - CER Instituto Medico /ID# 222193, Quilmes, Buenos Aires
  - Organizacion Medica de Investigacion (OMI) /ID# 222187, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - CIER Centro de Investigaciones en Enfermedades Reumaticas /ID# 231769, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto CAICI S.R.L /ID# 222191, Rosario, Santa Fe Province
  - CIMER Centro Integral de Medicina Respiratoria /ID# 222188, San Miguel de Tucumán, Tucumán Province
  - DOM Centro de Reumatologia /ID# 222194, Buenos Aires
  - Instituto Medico Strusberg /ID# 222189, Córdoba
  - Instituto de Cardiologia /ID# 226634, Santiago del Estero
- Australia (5):
  - Genesis Research Services /ID# 224060, Broadmeadow, New South Wales
  - BJC Health /ID# 223884, Paramatta, New South Wales
  - Private Practice - Scott Walter Graf /ID# 223958, Adelaide, South Australia
  - Emeritus Research /ID# 223883, Camberwell, Victoria
  - Joint West Rheumatology /ID# 223886, Murdoch, Western Australia
- Austria (6):
  - Klinikum Klagenfurt am Wörthersee /ID# 239628, Klagenfurt, Carinthia
  - Ordination Dr. Leeb /ID# 224293, Hollabrunn, Lower Austria
  - Dr. Georg Kurtz /ID# 225477, Gleisdorf, Styria
  - Dr. Maya Thun /ID# 224299, Vienna, Vienna
  - Ordination Doz. Grisar /ID# 224298, Vienna, Vienna
  - Rheuma-Zentrum Wien-Oberlaa GmbH /ID# 227853, Vienna, Vienna
- Belgium (14):
  - CHU Saint Pierre /ID# 223041, Brussels, Brussels Capital
  - Rhumaconsult SPRL /ID# 221825, Charleroi, Hainaut
  - Reuma Instituut Hasselt /ID# 221822, Hasselt, Limburg
  - Duplicate_CHU UCL Namur - site Godinne /ID# 222797, Godinne, Namur
  - Algemeen Stedelijk Ziekenhuis /ID# 224121, Aalst, Oost-Vlaanderen
  - Private practice Sint-Niklaas /ID# 224123, Sint-Niklaas, Oost-Vlaanderen
  - Onze Lieve Vrouw Hospital /ID# 223042, Aalst
  - AZ Sint-Jan Brugge /ID# 223713, Bruges
  - AZ Sint Lucas /ID# 223093, Bruges
  - Reumacentrum /ID# 222799, Genk
  - ReumaClinic /ID# 221353, Genk
  - Maertens, Gistel, BE /ID# 221823, Gistel
  - CHU de Liege /ID# 222201, Liège
  - AZ Alma Campus Sijsele /ID# 222214, Sijsele
- France (73):
  - Centre Hospitalier de Laon /ID# 224857, Laon, Aisne
  - Polyclinique saint Odilon /ID# 225576, Moulins, Allier
  - CH Cannes - les Broussailles /ID# 226160, Cannes, Alpes-Maritimes
  - CHU Strasbourg - Hopital de Hautepierre /ID# 222450, Strasbourg, Bas-Rhin
  - Hopital Saint Joseph /ID# 227221, Marseille, Bouches-du-Rhone
  - cabinet liberal- Dr CORNILLE /ID# 227869, Caen, Calvados
  - Centre Hospitalier d'Angouleme /ID# 226064, Angoulême, Charente
  - CHU Dijon /ID# 223799, Dijon, Cote-d Or
  - CH Georges Renon /ID# 225197, Niort, Deux-Sevres
  - CHU de Besancon - Jean Minjoz /ID# 222463, Besançon, Doubs
  - Cabinet de rhumatologie /ID# 227740, Mennecy, Essonne
  - Cabinet Rhumatologie St Michel Sur Orge /ID# 225176, Saint-Michel-sur-Orge, Essonne
  - Hopital de la Cavale Blanche /ID# 222462, Brest, Finistere
  - CH des Pays de Morlaix /ID# 223795, Morlaix, Finistere
  - CHU Limoges - Dupuytren 1 /ID# 222457, Limoges, Franche-Comte
  - CHU Bordeaux - Hopital Pellegrin /ID# 224837, Bordeaux, Gironde
  - CHU Toulouse - Hopital Purpan /ID# 223150, Toulouse, Haute-Garonne
  - CH Bigorre - Site de la Gespe /ID# 225141, Tarbes, Hautes-Pyrenees
  - CH Roubaix - Hopital Victor Provo /ID# 225032, Roubaix, Hauts-de-France
  - Clinique Beau Soleil /ID# 224238, Montpellier, Herault
  - CHU Montpellier - Hopital Saint Eloi /ID# 222452, Montpellier, Herault
  - CHU Montpellier - Hopital Saint Eloi /ID# 223394, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 223211, La Tronche, Isere
  - Cabinet médical /ID# 225000, Les Abrets En Dauphine, Isere
  - Cabinet médical /ID# 225321, Reims, Marne
  - Cabinet de Rhumatologie Poincare /ID# 224755, Thionville, Moselle
  - Cabinet liberal - Compiegne - Dr Banse /ID# 227099, Compiègne, Oise
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 222986, Paris, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 225787, Nantes, Pays de la Loire Region
  - CH Roanne /ID# 224729, Roanne, Pays de la Loire Region
  - CHU Nice -Hopital Pasteur /ID# 222460, Nice, Provence-Alpes-Côte d'Azur Region
  - Infirmerie Protestante /ID# 222438, Caluire-et-Cuire, Rhone
  - HCL - Hopital Lyon Sud /ID# 222447, Pierre-Bénite, Rhone
  - Cabinet medical /ID# 225366, Aix-les-Bains, Savoie
  - CHU Amiens-Picardie Site Sud /ID# 222444, Amiens, Somme
  - Cabinet libéral du Dr PAUPIERE /ID# 238723, Péronne, Somme
  - Cabinet medical /ID# 224850, Albi, Tarn
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 229086, La Roche-sur-Yon, Vendee
  - CH du Pays d'AIX /ID# 229561, Aix-en-Provence
  - Cabinet Novel d'Annecy /ID# 232310, Annecy
  - Centre Hospitalier d'Arras /ID# 223172, Arras
  - Centre Hospitalier de Boulogne Sur Mer /ID# 222991, Boulogne-sur-Mer
  - Centre Hospitalier Jean Rougie /ID# 224242, Cahors
  - CHRU Tours - Hopital Trousseau /ID# 222445, Chambray-lès-Tours
  - Centre Hospitalier de CHOLET /ID# 222455, Cholet
  - Hia Percy /Id# 225642, Clamart
  - CHU Clermont Ferrand - Hopital Gabriel Montpied /ID# 223801, Clermont-Ferrand
  - C. H. Sud Francilien /ID# 222446, Corbeil-Essonnes
  - Cabinet medical /ID# 225142, Haguenau
  - CH La Rochelle - Hopital Saint Louis /ID# 224240, La Rochelle
  - CH Emile Roux Le Puy en Velay /ID# 223688, Le Puy-en-Velay
  - CHU Lille - Hôpital Roger Salengro /ID# 223170, Lille
  - Clinique de la Sauvegarde /ID# 223424, Lyon
  - CH Princesse Grace /ID# 222451, Monaco
  - Ch Montauban /Id# 231854, Montauban
  - ELSAN - Clinique du Pont de Chaume /ID# 224898, Montauban
  - Ch Mulhouse /Id# 223442, Mulhouse
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 223591, Orléans
  - AP-HP - Hopital Saint-Antoine /ID# 222441, Paris
  - Hopital Pitie Salpetriere /ID# 222443, Paris
  - Cabinet medical /ID# 224855, Paris
  - Centre de Soins Osteoarticulaires Ambulatoires /ID# 224737, Paris
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 222449, Paris
  - GH Diaconesses Croix Saint-Simon /ID# 229126, Paris
  - CHU de Rennes - Hospital Sud /ID# 222458, Rennes
  - Clinique Saint-Hilaire /ID# 223833, Rouen
  - Hôpital Charles-Nicolle /ID# 223589, Rouen
  - Hôpital d'instruction des armées Bégin /ID# 222440, Saint-Mandé
  - CH Saint Nazaire /ID# 225750, Saint-Nazaire
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord /ID# 222456, Saint-Priest-en-Jarez
  - Cabinet rhumatologie Dr NECTOUX /ID# 225828, Sainte-Maxime
  - Groupe Médical Spécialisé - Le Premium /ID# 223719, Strasbourg
  - Hopital Avicenne - APHP /ID# 224248, Bobigny, Île-de-France Region
- Germany (19):
  - Praxis Dr. Haas /ID# 225187, Tübingen, Baden-Wurttemberg
  - Rheumatologische-Immunologische Praxis Templin /ID# 226924, Templin, Brandenburg
  - ACURA Rheumazentrum Baden-Bade /ID# 225225, Baden-Baden
  - Rheumapraxis Prof Dr Karin Manger /ID# 224086, Bamberg
  - Praxis fuer Rheumatologie und Innere Medizin /ID# 225222, Berlin
  - Eisterhues, Braunschweig, DE /ID# 225186, Braunschweig
  - Rheumatologie in Veedel /ID# 224999, Cologne
  - Dres. Karger/Baerlecken /ID# 224809, Cologne
  - Praxis Dilltal /ID# 226925, Ehringshausen
  - MVZ Ambulantes Rheumazentrum Erfurt /ID# 224812, Erfurt
  - Helios Fachklinik Vogelsang-Gommern /ID# 222949, Gommern
  - Asklepios MVZ Nord SH GmbH /ID# 225048, Hamburg
  - Heilig, Heidelberg, DE /ID# 225223, Heidelberg
  - Praxis internistische Rheumatologie /ID# 239226, Leipzig
  - Dres. Teipel/Toussaint/Saech /ID# 226923, Leverkusen
  - Aurich & Sieburg, Magdeburg /ID# 230701, Magdeburg
  - Die Fachaerzte im Rottal - Nephrologie, Rheumatologie /ID# 223866, Pfarrkirchen
  - MVZ für Rheumatologie Dr. M. Welcker /ID# 226926, Planegg
  - Krankenhaus der Barmherzigen Brüder Trier /ID# 226927, Trier
- Greece (13):
  - Olympion General Clinic /ID# 224130, Pátrai, Achaia
  - 251 Airforce General Hospital /ID# 225065, Athens, Attica
  - General Hospital of Athens Gennimatas /ID# 225064, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 224164, Athens, Attica
  - University General Hospital Attikon /ID# 224136, Athens, Attica
  - General Hospital Asklepieio Voulas /ID# 224131, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 224133, Heraklion, Crete
  - University General Hospital of Alexandroupolis /ID# 224880, Alexandroupoli, Evros
  - Naval Hospital of Athens /ID# 224135, Athens
  - General Hospital of Patras Agios Andreas /ID# 224132, Pátrai
  - Bioclinic Thessaloniki /ID# 224879, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 229965, Thessaloniki
  - Euromedica General Clinic /ID# 224134, Thessaloniki
- Ireland (4):
  - St James Hospital /ID# 224201, Dublin, Dublin
  - Hermitage Medical Clinic /ID# 239556, Dublin, Dublin
  - St Vincent's University Hospital /ID# 224200, Elm Park, Dublin
  - Tallaght University Hospital /ID# 231260, Tallaght, Dublin
- Israel (9):
  - Meir Medical Center /ID# 222116, Kfar Saba, Central District
  - HaEmek Medical Center /ID# 222138, Afula, H_efa
  - Hillel Yaffe Medical Center /ID# 222170, Hadera, H_efa
  - Rambam Health Care Campus /ID# 222118, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 223851, Haifa, H_efa
  - Galilee Medical Center /ID# 222113, Nahariya, Northern District
  - The Chaim Sheba Medical Center /ID# 222034, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 222117, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 222694, Haifa
- Italy (29):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Do Ancona /ID# 229440, Torette, Ancona
  - Azienda Ospedaliero Universitaria di Ferrara - Ospedale Sant'Anna /ID# 228788, Cona, Ferrara
  - ASL 3 Genovese - Ospedale la Colletta /ID# 228892, Arenzano, Genova
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 229061, Rome, Lazio
  - Ospedale San Raffaele IRCCS /ID# 229059, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 228807, Milan, Milano
  - Istituto Clinico Humanitas /ID# 227943, Rozzano, Milano
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 229063, Rome, Roma
  - Sapienza University /ID# 228014, Rome, Roma
  - Ospedale Mauriziano di Torino /ID# 228888, Turin, Torino
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo /ID# 228889, Alessandria
  - Azienda Ospedaliera Universitaria Consorziale Policlinico /ID# 228580, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni /ID# 228967, Bergamo
  - ASST Spedali civili di Brescia /ID# 228970, Brescia
  - Ospedale Ss. Annunziata /ID# 228809, Chieti
  - ASST Gaetano Pini/Presidio Ospedaliero Pini /ID# 228556, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 228554, Modena
  - AOU Universita degli Studi della Campania Luigi Vanvitelli /ID# 229057, Napoli
  - Ospedale San Giovanni Bosco /ID# 228552, Napoli
  - Azienda Ospedaliera Civico Di Cristina Benfratelli- P.O. Civico /ID# 228912, Palermo
  - Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 228160, Palermo
  - Fondazione IRCCS Policlinico /ID# 227937, Pavia
  - Azienda Ospedaliero Universitaria Pisana /ID# 228550, Pisa
  - Azienda Ospedaliera Regionale San Carlo /ID# 228648, Potenza
  - Azienda Ospedaliero-Universitaria Sant'Andrea /ID# 227942, Rome
  - Azienda Ospedaliera Universitaria "San Giovanni di Dio e Ruggi d'Aragona /ID# 229065, Salerno
  - Azienda Ospedaliero-Universitaria Senese-Ospedale Santa Maria delle Scotte /ID# 227938, Siena
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 228551, Udine
  - Azienda Ospedaliera Universitaria di Verona/Ospedale Borgo Trento /ID# 228553, Verona
- Kuwait (3):
  - Mubarak Hospital /ID# 224139, Hawalli
  - Ameeri Hospital /ID# 224140, Kuwait City
  - KOC Hospital /ID# 224138, Kuwait City
- Mexico (9):
  - Centro Integral en Reumatologia S.A de C.V /ID# 224363, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 224361, Guadalajara, Jalisco
  - Private Office Dr. Orozco /ID# 243257, Guadalajara, Jalisco
  - Centro de Estudios de Investigación Básica y Clínica, S.C. /ID# 224364, Guadalajara, Jalisco
  - RM Pharma Specialists S.A de C.V. /ID# 224359, Mexico City, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 240836, Mexico City, Mexico City
  - Consultorio Medico Privado - Miryam Eguia Bernal /Id# 243255, Monterrey, Nuevo León
  - Centro Especializado en Diabetes, Obesidad y Prevencion de Enfermedades Cardiova /ID# 224360, Mexico City
  - Consultorio Privado Jorge Rojas Serrano /Id# 243258, Puebla City
- Russia (18):
  - LLC MC RevmaMed /ID# 239162, Syktyvkar, Komi
  - Moscow Regional Research and Clinical Institute n.a. Vladimirskiy (MONIKI) /ID# 224852, Moscow, Moscow Oblast
  - Samara Regional Clinical Hospital n.a. V. D. Seredavin /ID# 227852, Samara, Samara Oblast
  - Nort-Western State Medical University n.a. Mechnikov /ID# 223419, Saint Petersburg, Sankt-Peterburg
  - GBUZ TO Regional Clinical Hospital No. 1 /ID# 241113, Tyumen, Tyumen Oblast
  - District clinical hospital /ID# 227662, Khanty-Mansyisk
  - City Clinical Hospital #52 /ID# 242947, Moscow
  - Omsk Regional Clinic Hospital /ID# 232029, Omsk
  - Orenburg State Medical University /ID# 243615, Orenburg
  - Republican hospital named after V.A. Baranov /ID# 227661, Petrozavodsk
  - Clinical Rheumatologic Hospital No 25 /ID# 242475, Saint Petersburg
  - Military Medical Academy n.a. Kirov /ID# 242351, Saint Petersburg
  - Clinic of Samara State Medical University /ID# 241168, Samara
  - Budgetary Institution of the Khanty-Mansiysk Autonomous Okrug-Yugra Surgut Dist /ID# 243313, Surgut
  - Nebbiolo Clinical Research Center /ID# 224900, Tomsk
  - Ulyanovsk Regional Clinical Hospital /ID# 239164, Ulyanovsk
  - Voronezh State Medical Univers /ID# 224854, Voronezh
  - Yaroslavl State Medicat University /ID# 224851, Yaroslavl
- Saudi Arabia (5):
  - Saudi German Hospital Jeddah /ID# 243234, Jeddah
  - King Abdulaziz University Hospital /ID# 222724, Jeddah
  - International Medical Center /ID# 243235, Jeddah
  - Saudi German Hospital /ID# 224137, Mushait
  - King Fahad Medical City /ID# 222917, Riyadh
- Spain (28):
  - Complejo Hospitalario Universitario A Coruña /ID# 231818, A Coruña, A Coruna
  - Hospital de Mérida /ID# 231826, Mérida, Badajoz
  - Hospital Universitari Mútua Terrassa /ID# 231822, Terrassa, Barcelona
  - Hospital de Viladecans /ID# 231823, Viladecans, Barcelona
  - Hospital Virgen del Puerto /ID# 240149, Plasencia, Caceres
  - Hospital Universitario de Jerez de la Frontera /ID# 231844, Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia /ID# 231843, Córdoba, Cordoba
  - Hospital Universitario de Getafe /ID# 231825, Getafe, Madrid
  - Hospital General Universitario Santa Lucia /ID# 238780, Cartagena, Murcia
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 231847, El Palmar, Murcia
  - Hospital Rafael Mendez /ID# 231846, Lorca, Murcia
  - Hospital Xeral Cies (CHUVI) /ID# 231819, Vigo, Pontevedra
  - Hospital Universitario Canarias /ID# 231848, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Ernest Lluch Martin /ID# 238779, Calatayud, Zaragoza
  - Hospital Universitario Torrecardenas /ID# 241931, Almería
  - Hospital Perpetuo Socorro /ID# 231827, Badajoz
  - Hospital Parc de Salut del Mar /ID# 240000, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 231821, Barcelona
  - Hospital General de Granollers /ID# 238778, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 231841, Granada
  - Hospital Juan Ramon Jimenez /ID# 231840, Huelva
  - Hospital Universitario de Jaen /ID# 231842, Jaén
  - Hospital Universitario Ramon y Cajal /ID# 241901, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 240150, Málaga
  - Hospital Universitario Virgen Macarena /ID# 231837, Seville
  - Hospital Universitario Virgen del Rocio /ID# 231836, Seville
  - Hospital Universitario Virgen de Valme /ID# 231838, Seville
  - Hospital Royo Villanova /ID# 231824, Zaragoza
- Switzerland (7):
  - Kantonsspital Aarau AG /ID# 222354, Aarau, Canton of Aargau
  - Universitätsspital Basel /ID# 224160, Basel Town, Canton of Basel-City
  - Kantonsspital St. Gallen /ID# 224158, Sankt Gallen, Canton of St. Gallen
  - CHUV, Centre hospitalier universitaire vaudois /ID# 224161, Lausanne, Canton of Vaud
  - Rheumatologisches Versorgungszentrum Weinfelden /ID# 222346, Weinfelden, Thurgau
  - Inselspital, Universitaetsspital Bern /ID# 224951, Bern
  - HFR Fribourg - Hôpital cantonal /ID# 224163, Fribourg
- Taiwan (6):
  - National Taiwan University Hospital /ID# 241050, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 241052, Kaohsiung City
  - China Medical University Hospital /ID# 241051, Taichung
  - Chi-Mei Medical Center /ID# 241745, Tainan
  - Tri-Service General Hospital /ID# 241746, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 241053, Taoyuan
- United Arab Emirates (4):
  - Cleveland Clinic Abu Dhabi /ID# 223176, Abu Dhabi
  - Integrated Rheumatology and Arthritis Center /ID# 223177, Dubai
  - Departnent of Medicine-Rheumatology Al Baraha Hospital and Al Qasmi Hospital Min /ID# 223178, Dubai
  - Drt Sulaiman Al Habib Hospital /ID# 226575, Dubai
- Uruguay (2):
  - Asociacion Española /ID# 222009, Montevideo
  - Medica Uruguaya /ID# 222008, Montevideo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ostor A, Feist E, Sidiropoulos P, Avouac J, Rebella M, Namas R, McDearmon-Blondell E, Gao T, Lagunes-Galindo I, Strengholt S, Zisman D, Attar S. Achievement of treatment targets and maintenance of response with upadacitinib in patients with moderate-to-severe rheumatoid arthritis in real-world practice: 1-year outcomes from the UPHOLD observational study. Arthritis Res Ther. 2025 Apr 10;27(1):84. doi: 10.1186/s13075-025-03528-5. PMID 40211417
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-095#additional-resources-section